CLINICAL TRIAL: NCT03243461
Title: International Cooperative Phase III Trial of the HIT-HGG Study Group for the Treatment of High Grade Glioma, Diffuse Intrinsic Pontine Glioma, and Gliomatosis Cerebri in Children and Adolescents < 18 Years.(HIT-HGG-2013)
Brief Title: International Cooperative Phase III Trial of the HIT-HGG Study Group (HIT-HGG-2013)
Acronym: HIT-HGG-2013
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Göttingen (Other)
Collaborators: Deutsche Kinderkrebsstiftung (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christof Kramm, Coordinating investigator, University of Göttingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01153; 2013-004187-56 (EudraCT Number)
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Glioblastoma WHO Grade IV; Diffuse Midline Glioma Histone 3 K27M WHO Grade IV; Anaplastic Astrocytoma WHO Grade III; Diffuse Intrinsic Pontine Glioma; Gliomatosis Cerebri
Keywords: Glioblastoma; high grade glioma; brain tumor; Anaplastic astrocytoma; DIPG; Gliomatosis cerebri; Diffuse midline glioma; Valproic acid; Temozolomide
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Neoplasms, Neuroepithelial; Glioblastoma; Glioma; Brain Neoplasms; Astrocytoma | interventions — Temozolomide; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temozolomide + Valproic acid (Experimental): E.g. Valproat-neuraxpharm®, Valproat-neuraxpharm® Lösung, Ergenyl®, Ergenyl®-Lösung oder Orfiril® Saft (Valproic acid), [10 mg/kg/d] tablet oder juice, p.o., every day in parallel to simultaneous radiochemotherapy with cytostatic drug Temodal (Temozolomid): [75 mg/m2/d] during simultaneous radiochemotherapy (7 days a week, max. 49 days); [150-200 mg/m2/d] during consolidation therapy (for 5 days every 28 days, 12 cycles), tablets, p.o. (or powder for preparation of an intravenously applicable solution).
  Interventions: Drug: Temozolomide + Valproic Acid

INTERVENTIONS:
Drug: Temozolomide + Valproic Acid — Valproic acid additionally to simultaneous radiochemotherapy with temozolomide

SUMMARY:
The HIT-HGG-2013 trial offers an innovative high-quality diagnostics and science program for children and adolescents >3 years, suffering from one of the following types of high grade gliomas:

1. glioblastoma WHO grade IV (GBM)
2. diffuse midlineglioma histone 3 K27M mutated WHO grade IV (DMG)
3. anaplastic astrocytoma WHO grade III (AA)
4. diffuse intrinsic pontine glioma (DIPG)
5. gliomatosis cerebri (GC) For 1.-3. diagnosis has to be confirmed by neuropathological survey, for 4. and 5. diagnosis has to be confirmed by neuroradiological survey.

In addition to standard treatment (radiotherapy and temozolomide chemotherapy) the effect of valproic acid which is traditionally used for treatment of seizure disorder, will be investigated. The aim of the trial will be to investigate whether this drug may increase the effects of radio- and chemotherapy, resulting in a better survival of the treated patients. Scientific studies provided evidence for anti-tumoral effects of valproic acid: the drug seems to be a so-called histondeacetylase inhibitor (HDAC inhibitor), controlling important genetic processes of tumor growth.

Studies in cell culture, animals and first clinical trials in adults as well provided evidence for efficacy of valproic acid in the treatment of glioblastoma. Due to this we hope children and adolescents suffering from GBM, DMG, AA, DIPG und GC will benefit from the treatment, too.

The aim of the HIT-HGG-2013 trial will be to compare the effects of Valproic acid with data of the HIT-HGG-2007 trial (children and adolescents with same diseases, only treated with simultaneous temozolomide radiochemotherapy).

In the present study, it was originally planned to investigate the therapeutic efficiency and safety of valproic acid and the autophagy inhibitor chloroquine, both in addition to temozolomide therapy. Since distribution of Resochin junior (chloroquine phosphate) was terminated, recruitment of new patients was stopped on August 8, 2019. For continuation of the trial, the chloroquine arm was closed but the patients already recruited in this arm will be followed up.

DETAILED DESCRIPTION:
Indication:

First-line treatment of high grade gliomas, diffuse intrinsic pontine glioma, and gliomatosis cerebri in paediatric patients < 18 years of age.

Background:

Based on published preclinical and clinical results regarding the potential therapeutic benefit of adult and pediatric high grade glioma patients receiving the histone deacetylase (HDAC) inhibitor valproic acid (VPA; Barker et al. 2013; Wolff et al. 2008, 2011; Felix et al. 2011; Su et al. 2011; Rokes et al. 2010; Masoudi et al. 2008; Guthrie et al. 2013; Weller et al. 2011) in addition to radiochemotherapy, the present trial is aimed to investigate if the addition of VPA to radiochemo- and maintenance therapy with temozolomide (Stupp et al. 2005; Cohen et al. 2011a, b) provides a survival advantage in comparison to radiochemo- and maintenance therapy with temozolomide alone. Therapeutic efficiency of VPA will be evaluated by comparison with a historical patient control from the previous trial HIT-HGG-2007 with temozolomide radiochemo- and maintenance therapy alone. Besides therapeutic efficiencies as indicated by event-free survival (EFS) and overall survival (OS) treatment-related toxicities will also be analysed.

Therapy:

TMZ and VPA will be studied as investigational medicinal products in the present trial.

* Trial treatment will be performed as follows: Surgery with best possible extent of tumour resection
* Start as soon as diagnosis is confirmed with VPA 10 mg/kg/d in two daily doses preferencially as NONRETARDED FORMULA (e.g. Valproat-neuraxpharm®, Valproat-neuraxpharm® Lösung, Ergenyl®, Ergenyl®-Lösung or Orfiril® Saft; however, any VPA preparation including generic drugs is allowed; the use of a retarded formula might be helpful in some case as indicated below), increase by 10 mg/kg/d once per week up until recommended target Serum level of 75-100 μg/ml (520-694 μmol/L) is reached. If target serum levels cannot be reached with non-retarded formula and/or side effects occur which might be connected to VPA, change to a retarded formula may be helpful to obtain sufficient VPA serum levels and/or reduce side effects. If VPA target serum levels are still not reached and/or side effects occur even with a retarded VPA formula, please contact the HIT-HGG study office.

After start of VPA induction with simultaneous radiochemotherapy:

* Fractionated, locoregional radiotherapy, total dose 54-60 Gy
* Simultaneous chemotherapy with oral temozolomide, 7 days per week at 75 mg/m2/d, starting at day 1 for the entire period of radiotherapy (at maximum 49 days; oral temozolomide treatment may be started in single cases at maximum 7 days before radiotherapy if the 49 days treatment period still fully covers radiotherapy).
* Please, use temozolomide capsules (for oral application) and temozolomide powder (for preparation of an intravenously applicable solution). Any temozolomide preparation including generic drugs is allowed except for patients who are not able to swallow capsules and in whom the use of an intravenous solution is no Option only Temodal® capsules must be used to generate a temozolomide suspension as described in the Appendix A.11. Parents have to be advised how to prepare the Temodal® suspension at the trial site. PLEASE NOTE: Capsules of generic temozolomide drugs other than Temodal® MUST NOT be opened and used for generating temozolomide suspension.
* Maintenance therapy with daily VPA and temozolomide four weeks after simultaneous radiochemotherapy initiation of a 5 day-course of oral temozolomide [150-200 mg/m2/d], repeated every 28 days for in total 12 courses VPA treatment is performed until day 28 of the 12th course of temozolomide.
* Treatment doses may vary according to available medication formulations and sizes. Thus, deviances of +/- 15% of the recommended doses may be acceptable if not stated otherwise.The starting points of treatment may also vary in single cases. Thus, deviances of +/- 7 days of the recommended time periods to start treatment may be acceptable if not stated otherwise.

Primary end point : Event-free survival

Biometry (regarding the primary objectives):

1. Confirmatory statistical design:

   1. Difference between the treatment with additional VPA and the historic sample from the HIT-HGG-2007 study with respect to EFS. Rejection of H0 will be interpreted as a significant difference between VPA treatment and the historic sample. A directional interpretation will detect either a superiority of the VPA-treatment compared to the historic sample, or a superiority of the historic sample compared to the VPA Treatment sample.

   Statistical tests: adaptive Log-rank test / (conventional) Log-rank test

   Multiple Significance level α(overall) = 5% Power = 80% Assumed 6 months EFS-rates = 55% vs. 70%

   Multiple Testing: No Multiplicity Problem in this trial.
2. Estimated sample sizes:

About 167 recruitments at final analysis

Patient recruitment will be performed for 5,4 years. Individual follow-up (including study treatment) is required for this protocol for at least 1 year and 30 days after study entry. Long-term follow-up is strongly recommended and will be organised according to national guidelines and recommendations.

Financial support:

Deutsche Kinderkrebsstiftung, Bonn, Germany

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, previously untreated diffuse paediatric high grade glioma with central neuropathological review including paedHGG (WHO grade IV) and anaplastic astrocytoma (WHO grade III).
* Newly diagnosed, previously untreated diffuse intrinsic pontine glioma with central neuroradiological review
* Newly diagnosed, previously untreated gliomatosis cerebri of all tumour grades with central neuroradiological review
* Patient ≥ 3 years and < 18 years of age at time of diagnosis
* Written informed consent of the patient and/or the patient's parents or legal guardian according to national laws

Exclusion Criteria:

* Pre-treatment of paedHGG (WHO grade IV), anaplastic astrocytoma (WHO grade III), diffuse intrinsic pontine glioma (as confirmed by neuroradiological review), and gliomatosis cerebri (as confirmed by neuroradiological review).
* Known hypersensitivity or contraindication to study drugs and/or dacarbazine
* Prior chemotherapy within the last 30 days before HIT-HGG-2013 treatment or radiotherapy which prevents adequate Performance of radiotherapy as outlined by the present protocol. This may mainly apply to patients with secondary high grade glioma after previous malignant brain tumour, e.g. medulloblastoma, ependymoma, craniopharyngeoma. If previous treatment does not prevent the adequate performance of the outlined Treatment protocol patients with secondary high grade glioma will be eligible for the present trial.
* Other (simultaneous) malignancies
* Pregnancy and / or lactation
* Patients who are sexually active refusing to use effective contraception (oral contraception, intrauterine devices, barrier method of contraception in conjunction with spermicidal jelly)
* Current or recent (within 30 days prior to start of trial treatment) treatment with another investigational drug or participation in another investigational trial.
* Clinical (e.g. a constitutional mismatch repair deficiency score ≥ 3; Wimmer et al. 2014) and/or other hints (e.g. absent intratumoral immunohistochemical expression of at least one of the MLH1, MSH2, MSH6, or PMS2 mismatch repair proteins and/or high microsatellite instability) for an underlying biallelic (constitutional) mismatch repair deficiency (bMMRD/CMMRD) or a heterozygous mismatch repair deficiency (hereditary non-polyposis colon cancer syndrome/HNPCC syndrome/Lynch syndrome): These patients and their relatives should be offered human genetic counseling and rapid genetic diagnostics to confirm or rule out These conditions. These patients might not benefit from the present study treatment but maybe from other therapeutic strategies (Bouffet et al. 2016). Since patients with clinically suspected neurofibromatosis type 1 may display similar symptoms as in CMMRD, patients with clinically suspected neurofibromatosis type 1 should be also checked for CMMRD as suggested above.
* Very poor clinical condition as defined by demand of mechanical ventilation and/or demand for intravenous catecholamines and/or very severe neurological damage equivalent to a coma and/or tetraplegia with complete incapability for communication (deafness, blindness, mutism)
* Severe concomitant diseases (e.g. immune deficiency syndrome; known tumour predisposition syndromes which do not affect adequate performance of the trial represent no exclusion criterion a priori
* Known HIV positivity
* Known severe manifest hepatic disease including hepatic porphyria as well as personal or family history of severe hepatic dysfunction, especially drug-related
* Known severe pancreatic disease
* Known lethal hepatic dysfunction in a sibling during valproic acid treatment
* Known urea cycle defect
* Known mitochondrial diseases caused by genetic mutations within the gene coding for the enzyme polymerase gamma (POLG), e.g. Alpers-Huttenlocher syndrome, as well as suspected POLGrelated disorders in children under the age of two years
* Known severe coagulation disorders (in regards to thrombopenia see prerequisite for blood cell count before starting treatment)
* Valproic acid as antiepileptc drug for any pre-existing epilepsy (Exception: Valproic acid treatment due to tumour-related epilepsy will be tolerated, if the time interval between start of valproic acid treatment and trial enrolment is ≤ 8 weeks.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 167 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of effects of valproine acid with respect to historical control group. | 5.4 years
  To confirm that the Event-Free Survival (EFS) in patients ≥ 3 years of age with paed HGG WHO grade IV, anaplastic astrocytoma WHO grade III (AAIII), DIPG, and gliomatosis cerebri differs for children treated with additional VPA compared to children in the historical HIT-HGG-2007 study sample.

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kramm, Prof., MD, Study Chair — University of Göttingen
Locations (51):
- Germany (51):
  - Universitätsklinik RWTH Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Charité Universitätsmedizin Berlin, Berlin
  - HELIOS Klinikum Berlin Buch, Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Kliniken der Stadt Köln gGmbH, Cologne
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Sana Kliniken Duisburg GmbH - Wedau Kliniken, Duisburg
  - HELIOS Klinikum Erfurt GmbH, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Angelika-Lautenschläger-Klinik, Heidelberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Gemeinschaftskrankenhaus Herdecke, Herdecke
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Gesundheit Nordhessen - Klinikum Kassel, Kassel
  - UKSH Kiel, Kiel
  - Gemeinschaftsklinikum Mittelrhein gGmbH, Koblenz
  - HELIOS Klinikum Krefeld, Krefeld
  - Universitätsklinikum Leipzig, Leipzig
  - UKSH Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg A. ö. R., Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - UMM Universitätsmedizin Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Technische Universität München / Klinikum Schwabing, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Universitäts-Kinder- und Jugendklinik Rostock, Rostock
  - ASKLEPIOS Klinik St. Augustin, Sankt Augustin
  - HELIOS Kliniken Schwerin GmbH, Schwerin
  - Klinikum Stuttgart - Olgahospital, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinik Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No